CLINICAL TRIAL: NCT03188575
Title: Digital IAPT: The Effectiveness & Cost-effectiveness of Internet-delivered Interventions for Depression and Anxiety Disorders in the Improving Access to Psychological Therapies Programme
Brief Title: Effectiveness & Cost-effectiveness of Internet-delivered Interventions for Depression and Anxiety Disorders in IAPT
Acronym: D-IAPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Silver Cloud Health (Other)
Collaborators: Berkshire Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-IAPT
Record Dates: First submitted 2017-06-08; First posted 2017-06-15 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Depression; Anxiety Disorders; Depressive Disorder; Generalized Anxiety Disorder; Social Anxiety Disorder; Phobic Disorders; Panic Disorder; Health Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders; Depressive Disorder; Generalized Anxiety Disorder; Phobia, Social; Phobic Disorders; Panic Disorder | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCBT for Depression and Anxiety (Experimental): SilverCloud Internet-Delivered Cognitive Behavioural Therapy
  Interventions: Behavioral: SilverCloud Internet-delivered Cognitive Behavioural Therapy
- Waiting List (Active Comparator): Waiting list control
  Interventions: Other: Waiting List

INTERVENTIONS:
Behavioral: SilverCloud Internet-delivered Cognitive Behavioural Therapy — SilverCloud Health is a leading provider of online therapeutic solutions to support and promote positive behavior change and mental wellness. SilverCloud delivers interventions for all of the anxiety disorders (panic disorder, social anxiety, phobias, GAD, health anxiety, OCD), depression and also comorbid depression and anxiety. The programs for the treatment of depression and anxiety employ several innovative engagement strategies for improving the user experience. These are divided into several categories: personal, interactive, supportive, and social. Research on the SilverCloud interventions has yielded significant clinical outcomes (Richards et al., 2015).
  Arms: iCBT for Depression and Anxiety
Other: Waiting List — 8 week waiting list period.
  Arms: Waiting List

SUMMARY:
Depression and anxiety are common mental health problems. There are effective treatments for depression and anxiety and one of these is talking therapies using cognitive behaviour therapy (CBT). In recent years CBT has been transferred to online delivery methods and these interventions have proven successful for people being treated with symptoms of depression and anxiety.

The current study will utilise a randomised controlled trial design, where the majority (n=240) of participants will be allocated to the immediate treatment (internet-delivered CBT for either depression or anxiety), and a smaller number (n=120) will be allocated to a waiting list. The waiting list group will receive treatment after an eight week wait. This design helps us to understand that any changes in symptoms in the treatment group will be likely due to the treatment they received compared to the waiting list.

A sample size of 360 participants is proposed and has been adjusted to ameliorate against patient dropout. Follow-up and maintenance of any positive changes in symptoms is very important in CBT for depression and anxiety, simply because some people can have a relapse of symptoms. We will therefore follow-up the treatment group for 3, 6, 9 and 12 months to assess maintenance of positive gains from treatment.

The study also seeks to investigate the cost effectiveness of the treatments.

DETAILED DESCRIPTION:
A CONSORT compliant single-blinded, parallel-groups, randomised controlled trial design will be used to examine the efficacy of internet-delivered interventions for depression and anxiety disorders against a waiting list control group. To be eligible participants will be screened and will need to score ≥ 9 on the PHQ-9 and / or ≥ 8 on the GAD-7. To establish a formal diagnosis of depression or anxiety, eligible participants will complete the M.I.N.I. neuropsychiatric interview and thereafter will be randomised to either an immediate treatment group or a waiting list group. Randomisation will follow a 2:1 ratio. The immediate treatment will complete a M.I.N.I. neuropsychiatric interview at 3-months follow-up from baseline. The treatment group will be followed up at 6-, 9- and 12-months post-treatment. The waiting list control group will be enrolled into the treatment once the immediate treatment group will have completed. The waiting list will complete baseline screening and research measures at baseline and similarly complete research measures at the end of the waiting period (8-weeks).

In addition, a nested study examining the mediators and moderators for change and maintenance of change is included. Specific and general mechanisms of change will be explored to include positive beliefs about repetitive negative thinking, therapeutic skills usage and therapist behaviours. General mediators including the therapeutic alliance and participant's expectancy / credibility and will be examined. The study protocol, information on the study, informed consent will be submitted for approval by the NHS England Research Ethics Committee and Health Research Authority approval for the study will be sought.

The study aims to evaluate the effectiveness and cost effectiveness of internet-delivered interventions for symptoms of depression and anxiety disorders in IAPT.

Individuals who contact Berkshire Healthcare NHS Foundation Trust to access IAPT psychological services will be eligible to participate. Recruitment will begin in May 2017 and will continue for 6 months until the numbers are reached or exceeded.

Using G-Power to calculate our sample size and based on a moderate between group effect size of d=0.5 with a power of 80% and a 2:1 randomisation procedure into immediate treatment for depression and/or anxiety and a corresponding waiting list control group returned a total sample of 288. Adding a 25% uplift to ameliorate against attrition gave a total sample size of 360. Therefore for depression a total sample of 120 in the treatment group and a corresponding 60 in the control group and the same ratio for anxiety disorders. The 2:1 randomisation procedure was implemented to reduce the concern of having many people waiting for treatment after presenting to the IAPT service.

PWP clinicians who are involved in the study trial as supporters to participants will be invited to take part in the research, to complete post-review alliance measures online, complete post review therapist behaviours checklist and volunteer for a semi-structured interview to collect qualitative data on therapeutic alliance and therapist behaviours.

ELIGIBILITY:
Inclusion Criteria:

1. A score of ≥ 9 on PHQ-9 and/ or a score of ≥ 8 on GAD-7
2. 18 years of age
3. Suitable for an internet-delivered intervention (iCBT)

Exclusion Criteria:

1. Suicidal intent/ideation
2. Psychotic illness
3. Currently in psychological treatment for depression and/or anxiety
4. Alcohol or drug misuse
5. Previous diagnosis of an organic mental health disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-07-25 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Depression symptoms | Baseline, at treatment review sessions (maximum of 6 across an 8 week treatment period), 8 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up and 12 month follow-up
  Measured by the 9 item Patient Health Questionnaire (PHQ-9)
Change in Anxiety symptoms | Baseline, at treatment review sessions (maximum of 6 across an 8 week treatment period), 8 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up and 12 month follow-up
  Measured by the 7 item Generalised Anxiety Disorder inventory (GAD-7)

SECONDARY OUTCOMES:
Work and Social Adjustment | Baseline, at treatment review sessions (maximum of 6 across an 8 week treatment period), 8 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up and 12 month follow-up
  Measured using the Work and Social Adjustment scale (WSAS)
Social Anxiety | Baseline, at treatment review sessions (maximum of 6 across an 8 week treatment period), 8 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up and 12 month follow-up
  Measured using the Social Phobia Inventory (SPIN)
Health Anxiety | Baseline, at treatment review sessions (maximum of 6 across an 8 week treatment period), 8 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up and 12 month follow-up
  Measured using the Short Health Anxiety Inventory (SHAI)
Panic | Baseline, at treatment review sessions (maximum of 6 across an 8 week treatment period), 8 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up and 12 month follow-up
  Measured using the Panic Disorder Severity Scale (PDSS)
Generalised Anxiety Symptoms | Baseline, at treatment review sessions (maximum of 6 across an 8 week treatment period), 8 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up and 12 month follow-up
  Measured using the Penn State Worry Questionnaire (PSWQ)
Quality of life | baseline, 8 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up and 12 month follow-up
  Measured using the EQ5D5L
Quality of life for users of mental health services | baseline, 8 weeks, 3 month follow-up, 6 month follow-up, 9 month follow-up and 12 month follow-up
  Measured using the Re-QOL
Client service usage | baseline, 8 weeks, 6 month follow-up, 9 month follow-up and 12 month follow-up
  Measured using the Client Services Receipt Inventory (CSRI)
Emotion Regulation | Baseline and 8 weeks
  Measured using the Emotion Regulation Questionnaire (ERQ)
Rumination | Baseline and 8 weeks
  Measured using the Positive Beliefs about Depressive Rumination scale (PBRS-A)
Therapeutic Expectancy | Baseline, 4 weeks and 8 weeks.
  Measured using the Expectancy/Credibility scale (TEQ)
CBT Skills Usage | 3 month follow-up, 6 month follow-up, 9 month follow-up and 12 month follow-up
  Measured using the Frequency of Actions and Thoughts scale (FATS)
Therapist Behaviours | Continuous during treatment after each session for 8 weeks
  Measured using the Therapist Behaviours Checklist (TBCL)
Therapeutic Alliance for patients | Continuous during treatment after each session for 8 weeks
  Measured using the Scale to Assess Therapeutic Relationships - Patient Version (STAR-P)
Therapeutic Alliance for clinicians | Continuous during treatment after each session for 8 weeks
  Measured using the Scale to Assess Therapeutic Relationships - Clinician version (STAR-C)
Therapeutic Alliance for clinicians | During the patient recruitment period.
  Semi-structured interview will be employed to assess qualitatively clinicians experience of the therapeutic relationship online.
M.I.N.I. International Neuropsychiatric Interview | Baseline and 3-month follow-up
  Used to determine a diagnosis of depression and/or anxiety (MINI)
Patient Experience/Satisfaction | Post treatment (up to 8 weeks).
  Measured using the Patient Experience Questionnaire (PEQ)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Richards, PhD, Study Director — SilverCloud Health; Sarah Sollesse, MSc, Principal Investigator — Berkshire Healthcare NHS Foundation Trust
Locations (1):
- Berkshire NHS Foundation Trust, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Available on request from the PI

REFERENCES:
- [Background] Richards D, Timulak L, O'Brien E, Hayes C, Vigano N, Sharry J, Doherty G. A randomized controlled trial of an internet-delivered treatment: Its potential as a low-intensity community intervention for adults with symptoms of depression. Behav Res Ther. 2015 Dec;75:20-31. doi: 10.1016/j.brat.2015.10.005. Epub 2015 Oct 21. PMID 26523885
- [Derived] Richards D, Duffy D, Blackburn B, Earley C, Enrique A, Palacios J, Franklin M, Clarke G, Sollesse S, Connell S, Timulak L. Digital IAPT: the effectiveness & cost-effectiveness of internet-delivered interventions for depression and anxiety disorders in the Improving Access to Psychological Therapies programme: study protocol for a randomised control trial. BMC Psychiatry. 2018 Mar 2;18(1):59. doi: 10.1186/s12888-018-1639-5. PMID 29499675